CLINICAL TRIAL: NCT00647452
Title: Very Low Density Lipoprotein (VLDL) Triglyceride Metabolism in Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ES-0002
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Lipid metabolism; VLDL; Exercise; Lipid metabolism in exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Healthy male volunteers
  Interventions: Behavioral: Exercise
- 2 (Experimental): Healthy female volunteers
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate Intensity Exercise (50 % af VO2max) for 90 minutes

SUMMARY:
Purpose:

To investigate VLDL-TG metabolism in exercise in healthy volunteers to determine the contribution of VLDL-TG in exercise and eventual gender differences

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age: 20-50 years
* Premenopausal

Exclusion Criteria:

* Smoking
* Alcohol abuse
* Use of medications

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
VLDL-TG turnover | Hours

CONTACTS AND LOCATIONS:
Overall Officials: Esben Søndergaard, M.D., Principal Investigator — Medical Department M
Locations (1):
- Department of Endocrinology M, Aarhus Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] Mittendorfer B, Horowitz JF, Klein S. Effect of gender on lipid kinetics during endurance exercise of moderate intensity in untrained subjects. Am J Physiol Endocrinol Metab. 2002 Jul;283(1):E58-65. doi: 10.1152/ajpendo.00504.2001. PMID 12067843
- [Background] Gormsen LC, Jensen MD, Nielsen S. Measuring VLDL-triglyceride turnover in humans using ex vivo-prepared VLDL tracer. J Lipid Res. 2006 Jan;47(1):99-106. doi: 10.1194/jlr.M500205-JLR200. Epub 2005 Oct 18. PMID 16234572